CLINICAL TRIAL: NCT06692062
Title: A Prospective Study of Hypofractionated Radiotherapy for Thymic Epithelial Tumors
Brief Title: Hypofractionated Radiotherapy for Thymic Epithelial Tumors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rongrong Zhou (Other)
Responsible Party: Sponsor-Investigator, Rongrong Zhou, Deputy Director of Department of Oncology, Xiangya Hospital of Central South University
Organization: Xiangya Hospital of Central South University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202401009
Record Dates: First submitted 2024-11-13; First posted 2024-11-18 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Thymoma and Thymic Carcinoma; Thymoma; Thymic Cancer; Thymic Epithelial Tumor
Keywords: thymoma; hypofractionated radiotherapy; thymic carcinoma
MeSH Terms: conditions — Thymoma; Thymus Neoplasms; Thymic epithelial tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hypofractionated Radiotherapy (Experimental): R0 resection: 42-48 Gy/14-16f or 40-44 Gy or 10-11f,40 Gy/8f R1 resection: 48-51 Gy/16-17f or 44-48 Gy/11-12f or 40-45 Gy/8-9f R2 resection: 51-60 Gy/17-20f or 48-56 Gy/12-14f or 45 -60Gy/9-12f
  Interventions: Radiation: Hypofractionated Radiation Therapy
- Conventional Radiotherapy (No Intervention): R0 resection: 45-50Gy/20-25f R1 resection: 54-56Gy/25-28f R2 resection: 60-70Gy/30-35f

INTERVENTIONS:
Radiation: Hypofractionated Radiation Therapy — R0 resection: 45-50Gy/20-25f R1 resection: 54-56Gy/25-28f R2 resection: 60-70Gy/30-35f
  Arms: Hypofractionated Radiotherapy

SUMMARY:
The goal of this clinical trial is to learn if hypofractionated radiotherapy works to shorten the treatment time without increasing the side effects in patients of thymic epithelial tumors. The main questions it aims to answer are:

* Does Hypofractionated radiotherapy provide better results?
* Can hypofractionated radiotherapy reduce toxic and side effects compared with conventional radiotherapy? Researchers will compare the efficacy and safety of hypofractionated radiotherapy after thymic tumor surgery.

Participants will:

* Receive hypofractionated radiotherapy or conventional radiotherapy
* Visit the hospital regularly once every 12 weeks for checkups and tests

DETAILED DESCRIPTION:
According to the World Health Organization histological classification system, thymic epithelial tumors (TET) are divided into thymoma and thymic carcinoma. Surgery is the main treatment for thymic tumors, and radiotherapy (RT), as an important auxiliary method of surgery, also plays an irreplaceable role in all stages of thymoma.

Hypofractionated radiotherapy is a common mode of radiotherapy for thoracic tumors. Unlike conventional radiotherapy, hypofractionated radiotherapy has a higher single dose and a shorter course of treatment. Because it improves the treatment efficiency, it can reduce the treatment time of patients and medical institutions and the cost of patients.

In the postoperative radiotherapy stage, conventional radiotherapy and hypofractionated radiotherapy were used. The course of hypofractionated radiotherapy was shorter than that of conventional radiotherapy. Patients chose to accept hypofractionated radiotherapy as the hypofractionated group, but not the conventional group.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must provide written informed consent.
2. 18 years old ≤ age <75 years old.
3. Thymoma confirmed by pathology: type A, type AB, type B1, type B2, type B3. Thymic carcinoma. Patients with previous thymectomy were required to have complete surgical related data.
4. Masaoka⁃Koga ⁃ stage Ⅰ-Ⅲ
5. ECOG performance status 0-2.
6. Expected survival time > 1 year.
7. Participants of childbearing age must agree to use effective contraception during the trial; In women of childbearing age, a serum or urine pregnancy test must be negative.
8. Patients who are not lactating.
9. Sufficient bone marrow reserve and good function of important organs.

Exclusion Criteria:

1. patients with prior thoracic radiotherapy;
2. diseases not suitable for radiotherapy, such as recent myocardial infarction, active congestive heart failure;
3. Uncontrolled infectious disease or other serious medical or mental illness that may interfere with care
4. Patients with other malignant tumors that are not under stable control;
5. Known history of mental illness, substance abuse, alcohol or drug abuse.
6. Other conditions deemed unsuitable for enrollment by the attending physician.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2027-11-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
3-year PFS | The patients were followed up for 3 years from enrollment to disease progression or death.
  Time from enrollment to disease progression or death.

SECONDARY OUTCOMES:
toxicity | Patients were followed from enrollment until 3 years.
  Any adverse medical event that occurred between the time the patient provided informed consent and was enrolled in the trial and the date of the last follow-up visit.
3-year OS | The patients were followed up for 3 years from enrollment to death.
  Time from patient enrollment to patient death.

CONTACTS AND LOCATIONS:
Locations (1):
- Xiangya Hospital, Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No